CLINICAL TRIAL: NCT05472571
Title: FOREST HEALTH: Pilot Project of Forest Bathing for Promoting Health, Human Wellbeing, and for Complementing Sustainable Management Forest and Landscape Practices
Brief Title: Pilot Project of Forest Bathing for Promoting Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Collaborators: La Caixa Foundation (Other); Fundación Caja Navarra (Unknown)
Responsible Party: Principal Investigator, Ana Villarroya, Associate Professor, Clinica Universidad de Navarra, Universidad de Navarra
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BOSQUE
Record Dates: First submitted 2022-07-19; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Intellectual Disability
MeSH Terms: conditions — Intellectual Disability | interventions — Forest Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Forest bathing (Experimental)
  Interventions: Other: Forest bathing

INTERVENTIONS:
Other: Forest bathing — The intervention consists of 11 consecutive sessions of forest bathing (one session per week), each one lasting about 2 hours. Each session involves an easy walk through a forest area, interspersed with non-intrusive activities of contact with the surrounding nature aimed at fostering mindfulness and the use of the five senses.

SUMMARY:
An exploratory trial using a cuasi-experimental design aimed to improve the quality of life of people with intellectual disabilities. The intervention consists of 11 consecutive sessions of forest bathing (one session per week), each one lasting about 2 hours. Each session involves an easy walk through a forest area, interspersed with non-intrusive activities of contact with the surrounding nature aimed at fostering mindfulness and the use of the five senses. Data were collected at baseline, post intervention, and 7 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adults with intellectual disability enrolled in a specific occupational center.
* Being informed about the study and having signed the informed consent document.

Exclusion Criteria:

* Having stated their not willing to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Systolic and diastolic blood pressure | 1 minute
Heart coherence | 5 minutes
  Using emWave Pro Plus device and software
Perceived quality of life and wellbeing | 30 minutes
  Using INICO-FEAPS questionnaire (Verdugo Alonso et al., 2013): Scale for the Integral Evaluation of the Quality of Life of people with intellectual or developmental disability, developed by the University Institute for Community Integration (INICO) and the Spanish Confederation of Organizations for People with Intellectual or Developmental Disability (FEAPS).
  It is a self-report tool that consists of 72 four-point Likert-type items divided among 8 dimensions: self-determination, rights, emotional wellbeing, social inclusion, personal development, interpersonal relationships, material well-being, and physical well-being. Each dimension is composed of nine items. Each subscale score is calculated by summing up the score for each of the nine items, and a total score is then calculated by summing up the scale scores. Higher scores are associated to better quality of life.

SECONDARY OUTCOMES:
Physiological Equivalent Temperature | 10 minutes
  Following Höppe (1999) procedure
Thermic perception | 3 minutes
  Using questionnaire published in previous studies (Teli et al., 2012; Trebilcock et al., 2017), that includes 3 items to assess thermal sensation vote (TMV) (7-point Likert scale), one item to assess thermal preference vote (TPV) (3-point scale), one item to assess the feeling of comfort (closed-answer), one item to get clothing information (closed-answer), and one item to evaluate the feeling of tiredness (3-point scale). The answers to these questions put the PET value (outcome 4) into context and help interpret it.
Barriers and facilitators | 2 hours
  Field diary

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Navarra, Pamplona, Navarre, Spain

REFERENCES:
- [Background] Hoppe P. The physiological equivalent temperature - a universal index for the biometeorological assessment of the thermal environment. Int J Biometeorol. 1999 Oct;43(2):71-5. doi: 10.1007/s004840050118. PMID 10552310